CLINICAL TRIAL: NCT02270463
Title: A Phase 1/2 Study of SL-401 as Consolidation Therapy for Adult Patients With Adverse Risk Acute Myeloid Leukemia in First CR, and/or Evidence of Minimal Residual Disease (MRD) in First CR
Brief Title: SL-401 as Consolidation Therapy in Patients With Adverse Risk Acute Myeloid Leukemia in First Complete Remission
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STML-401-0214
Record Dates: First submitted 2014-10-09; First posted 2014-10-21 (Estimated); Results first posted 2024-08-21 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — tagraxofusp

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tagraxofusp-erzs (Experimental): Patients received tagraxofusp-erzs (SL-401) by IV infusion over 15 minutes for 5 consecutive days of a 28-day cycle in both stages.
  Interventions: Drug: Tagraxofusp-erzs

INTERVENTIONS:
Drug: Tagraxofusp-erzs — Tagraxofusp-Erzs administered by IV infusion at doses of 7, 9, and 12 µg/kg/day
  Other Names: SL-401

SUMMARY:
This is a non-randomized, open-label, multicenter, dose escalation study designed to determine the maximum tolerated dose (MTD) of SL-401 in adult patients with acute myeloid leukemia, and to evaluate the safety profile of SL-401 at the MTD.

DETAILED DESCRIPTION:
Patients who were in their first or second complete remission (CR) or complete remission with incomplete bone marrow recovery (CRi) after induction therapy were treated with SL-401, which was administered as a brief intravenous infusion for 5 consecutive days every 28 days for 6 or more cycles. Stage 1 consisted of a period in which patients were treated with SL-401 at 3 dose levels. During Stage 2, patients with minimal residual disease (MRD) in their bone marrow were treated at a MTD or maximum tested dose in which multiple dose-limiting toxicities were not observed (identified in Stage 1).

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a diagnosis of AML according to World Health Organization (WHO) criteria.
2. The patient received any induction chemotherapy regimen and may have received post-remission consolidation therapy prior to screening.
3. The patient has achieved a first or second CR or CRi. For patients without evidence of MRD in CR/CRi, CR (or CRi) must have been initially identified within 12 months prior to screening.

   OR The patient has achieved first or second CR or CRi with evidence of MRD as determined locally at least 6 months post stem cell transplant without evidence of acute or chronic graft-versus-host disease post-transplant and has not received immunosuppressant therapy for at least 14 days prior to SL-401 therapy.
4. The patient has adverse risk disease or AML for which there is otherwise a substantial risk of relapse, which includes but is not limited to: adverse karyotype, FLT3 internal tandem duplication (ITD) mutation, history of antecedent hematologic disorder (AHD), therapy-related AML, history of requiring more than 1 cycle of intensive induction chemotherapy to achieve first remission, and/or presence of persistent MRD (detected by cytogenetics, molecular markers, or flow cytometry) at any point after the initial induction cycle.
5. For patients enrolling in Stage 2, the bone marrow evaluation determined locally within the previous 6 months indicates the presence of MRD.
6. The patient is not considered to be an immediate candidate for allogeneic stem cell transplant as determined by the investigator.
7. The patient is ≥18 years old.
8. The patient has an Eastern Cooperative Oncology Group (ECOG) performance score (PS) of 0-2.
9. The patient has adequate organ function, including cardiac, renal, and hepatic function:

   * Left ventricular ejection fraction (LVEF) ≥institutional lower limit of normal as measured by multigated acquisition scan (MUGA) or 2-dimensional (2-D) echocardiography (ECHO) within 28 days prior to start of therapy and no clinically significant abnormalities on a 12-lead electrocardiogram (ECG)
   * Serum creatinine ≤1.5 mg/dL
   * Serum albumin ≥3.2 g/dL in the absence of receipt of (IV) albumin within the previous 72 hours.
   * Bilirubin ≤1.5 mg/dL
   * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 × the upper limit of normal (ULN)
   * Creatine phosphokinase (CPK) ≤2.5 × the ULN.
10. The patient has adequate bone marrow reserve:

    • Absolute neutrophil count (ANC) > 0.5 × 10^9/L
11. The patient is a woman of child bearing potential (WOCBP) who has had a negative serum or urine pregnancy test within 1 week prior to SL-401 treatment (intervals shorter than 1 week are acceptable if required by institutional guidelines).
12. A written and voluntarily signed informed consent must be obtained from the patient or legally authorized representative, in accordance with local regulations, before the initiation of any study related procedures. The patient or legally authorized representative must be able to read and understand the informed consent form (ICF).
13. The patient is able to adhere to the study visit schedule and other protocol requirements, including follow-up for survival assessment.
14. The patient (male and female) agrees to use acceptable contraceptive methods for the duration of time on the study, and continue to use acceptable contraceptive methods for 2 months after the last infusion of SL-401.

Exclusion Criteria:

1. The patient has a diagnosis of AML associated with karyotype t(15;17).
2. The patient has persistent and clinically significant Grade ≥2 toxicities from induction or consolidation therapy (excluding alopecia, nausea, fatigue, and liver function tests [as mandated in the inclusion criteria]) not readily managed with supportive measures.
3. The patient received treatment with another investigational agent within 14 days of screening.
4. The patient previously received treatment with SL-401.
5. The patient has an active malignancy and/or cancer history (excluding AML or antecedent myelodysplastic syndrome [MDS]) that may confound the assessment of the study endpoints. Patients with a past cancer history (within 2 years of entry) with substantial potential for recurrence and/or ongoing active malignancy must be discussed with the Sponsor before study entry. Patients with the following neoplastic diagnoses are eligible: non-melanoma skin cancer, carcinoma in situ, cervical intraepithelial neoplasia, organ-confined prostate cancer with no evidence of progressive disease.
6. The patient has clinically significant cardiovascular disease (e.g., uncontrolled or any New York Heart Association [NYHA] Class 3 or 4 congestive heart failure, uncontrolled angina, history of myocardial infarction, unstable angina or stroke within 6 months prior to study entry, uncontrolled hypertension or clinically significant arrhythmias not controlled by medication).
7. The patient has uncontrolled, clinically significant pulmonary disease (e.g., chronic obstructive pulmonary disease, pulmonary hypertension) that in the opinion of the Investigator would put the patient at significant risk for pulmonary complications during the study.
8. The patient has known active or suspected central nervous system (CNS) leukemia. If suspected, CNS leukemia should be ruled out with relevant imaging and/or examination of cerebrospinal fluid.
9. The patient has uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, disseminated intravascular coagulation (DIC), or psychiatric illness/social situations that would limit compliance with study requirements.
10. The patient is pregnant or breast feeding.
11. The patient has known positive status for human immunodeficiency virus (HIV), active or chronic Hepatitis B or Hepatitis C.
12. The patient is oxygen-dependent.
13. The patient has any medical condition which in the opinion of the Investigator places the patient at an unacceptably high risk for toxicities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Albert Einstein College of Medicine, The Bronx, New York
  - Tennessee Oncology, Nashville, Tennessee
  - M.D. Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Institute, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 1: Tagraxofusp-erzs 7 μg/kg/Day: Tagraxofusp-erzs (SL-401) 7 μg/kg/day by IV infusion over 15 minutes for 5 consecutive days of a 28-day cycle.
- Stage 1: Tagraxofusp-erzs 9 μg/kg/Day: Tagraxofusp-erzs (SL-401) 9 μg/kg/day by IV infusion over 15 minutes for 5 consecutive days of a 28-day cycle.
- Stage 1: Tagraxofusp-erzs 12 μg/kg/Day; Stage 2: Tagraxofusp-erzs 12 μg/kg/Day: Tagraxofusp-erzs (SL-401) 12 μg/kg/day by IV infusion over 15 minutes for 5 consecutive days of a 28-day cycle.
Period: Overall Study
Arm/Group | Stage 1: Tagraxofusp-erzs 7 μg/kg/Day | Stage 1: Tagraxofusp-erzs 9 μg/kg/Day | Stage 1: Tagraxofusp-erzs 12 μg/kg/Day | Stage 2: Tagraxofusp-erzs 12 μg/kg/Day
Started | 3 | 3 | 3 | 7
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Stage 1: Tagraxofusp-erzs 9 μg/kg/Day: Tagraxofusp-erzs (SL-401) 7 μg/kg/day by IV infusion over 15 minutes for 5 consecutive days of a 28-day cycle
- Total: Total of all reporting groups
Arm/Group | Stage 1: Tagraxofusp-erzs 7 μg/kg/Day | Stage 1: Tagraxofusp-erzs 9 μg/kg/Day | Stage 1: Tagraxofusp-erzs 12 μg/kg/Day | Stage 2: Tagraxofusp-erzs 12 μg/kg/Day | Total
Number analyzed (Participants) | 3 | 3 | 3 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (7.00) | 66.3 (10.69) | 59.0 (7.00) | 63.9 (14.02) | 63.8 (10.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 6 | 7
  Male | 2 | 3 | 3 | 1 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 3 | 3 | 6 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 3 | 2 | 3 | 6 | 14
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Dose-Limiting Toxicity (DLT)
Description: The maximum tolerated dose was defined as the dose preceding the dose level at which 2 or more patients experienced a DLT during treatment Cycle 1.
Time Frame: 24 weeks
Measure: Number; unit: events
Groups:
- Stage 1: Tagraxofusp-erzs 7 µg/kg/Day: Patients received tagraxofusp-erzs (SL-401) 7 µg/kg/day by IV infusion over 15 minutes for 5 consecutive days of a 28-day cycle in the absence of disease progression or other withdrawal criteria.
- Stage 1: Tagraxofusp-erzs 9 µg/kg/Day: Patients received tagraxofusp-erzs (SL-401) 9 µg/kg/day by IV infusion over 15 minutes for 5 consecutive days of a 28-day cycle in the absence of disease progression or other withdrawal criteria.
- Stage 1: Tagraxofusp-erzs 12 µg/kg/Day; Stage 2: Tagraxofusp-erzs 12 µg/kg/Day: Patients received tagraxofusp-erzs (SL-401) 12 µg/kg/day by IV infusion over 15 minutes for 5 consecutive days of a 28-day cycle in the absence of disease progression or other withdrawal criteria.
Arm/Group | Stage 1: Tagraxofusp-erzs 7 µg/kg/Day | Stage 1: Tagraxofusp-erzs 9 µg/kg/Day | Stage 1: Tagraxofusp-erzs 12 µg/kg/Day | Stage 2: Tagraxofusp-erzs 12 µg/kg/Day
Number analyzed (Participants) | 3 | 3 | 3 | 7
events | 0 | 0 | 0 | 0

2. Secondary Outcome: Eradication of Minimal Residual Disease (MRD) From Baseline
Description: The rate of MRD eradication (conversion) is defined as the proportion of patients with evidence of MRD prior to initial therapy with investigational SL-401 for whom MRD cannot be detected upon subsequent (post treatment) assessments.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Stage 2: Tagraxofusp-erzs 12 μg/kg/Day: Patients received tagraxofusp-erzs (SL-401) 12 μg/kg/day by IV infusion over 15 minutes for 5 consecutive days of a 28-day cycle in the absence of disease progression or other withdrawal criteria.
Arm/Group | Stage 1: Tagraxofusp-erzs 7 µg/kg/Day | Stage 1: Tagraxofusp-erzs 9 µg/kg/Day | Stage 1: Tagraxofusp-erzs 12 µg/kg/Day | Stage 2: Tagraxofusp-erzs 12 μg/kg/Day
Number analyzed (Participants) | 3 | 3 | 3 | 7
Participants
  MRD at Baseline | 1 | 2 | 1 | 5
  MRD Eradicated at Single Assessment | 1 | 1 | 0 | 0
  MRD Eradicated at Multiple Assessments | 0 | 1 | 0 | 0

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of first infusion of SL-401 to the date of death from any cause. Participants still alive or lost to follow-up at the time of analysis were censored on the last date known to be alive prior to the analysis cutoff date, as determined by in-person visit or telephone contact.
Time Frame: Day 1 (enrollment) through Month 44
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stage 1: Tagraxofusp-erzs 7 µg/kg/Day | Stage 1: Tagraxofusp-erzs 9 µg/kg/Day | Stage 1: Tagraxofusp-erzs 12 µg/kg/Day | Stage 2: Tagraxofusp-erzs 12 µg/kg/Day
Number analyzed (Participants) | 3 | 3 | 3 | 7
months | 12.2 [5.4 to NA] — Values were non-estimable (insufficient number of participants with events). | 21.9 [2.6 to NA] — Values were non-estimable (insufficient number of participants with events). | 19.0 [NA to NA] — Values were non-estimable (insufficient number of participants with events). A median value is reported only since the survival curve crossed 0.5 probability. Only 1 participant experienced the event. The other 2 participants were censored due to a shorter OS duration. | NA [5.9 to NA] — Values were non-estimable (insufficient number of participants with events).

4. Secondary Outcome: Relapse-Free Survival (RFS)
Description: RFS is defined as the proportion of patients who remain free of acute myeloid leukemia recurrence (hematologic) and alive.
Time Frame: 24 weeks
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Stage 1: Tagraxofusp-erzs 7µg/kg/Day: Patients received tagraxofusp-erzs (SL-401) 7 µg/kg/day by IV infusion over 15 minutes for 5 consecutive days of a 28-day cycle in the absence of disease progression or other withdrawal criteria.
Arm/Group | Stage 1: Tagraxofusp-erzs 7µg/kg/Day | Stage 1: Tagraxofusp-erzs 9 µg/kg/Day | Stage 1: Tagraxofusp-erzs 12 µg/kg/Day | Stage 2: Tagraxofusp-erzs 12 µg/kg/Day
Number analyzed (Participants) | 3 | 3 | 3 | 7
months | 2.7 [0.5 to NA] — Values were non-estimable (insufficient number of participants with events). | 5.1 [0.5 to NA] — Values were non-estimable (insufficient number of participants with events). | 5.4 [3.0 to NA] — Values were non-estimable (insufficient number of participants with events). | 5.0 [1.8 to 8.7]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed for up to 266 days. All-Cause Mortality was assessed for up to 44 months.
Description: An AE is any untoward medical occurrence in a study patient who is administered a medicinal product (drug or biologic); the event may or may not have a causal relationship with the medicinal product.
Groups:
- Stage 1: Tagraxofusp-erzs 9 µg/kg/da: Patients received tagraxofusp-erzs (SL-401) 9 µg/kg/day by IV infusion over 15 minutes for 5 consecutive days of a 28-day cycle in the absence of disease progression or other withdrawal criteria.
Arm/Group | Stage 1: Tagraxofusp-erzs 7 µg/kg/Day | Stage 1: Tagraxofusp-erzs 9 µg/kg/da | Stage 1: Tagraxofusp-erzs 12 µg/kg/Day | Stage 2: Tagraxofusp-erzs 12 µg/kg/Day
All-Cause Mortality (participants affected / at risk) | 3/3 | 2/3 | 1/3 | 3/7
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 3/3 | 4/7
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: Tagraxofusp-erzs 7 µg/kg/Day (N=3) | Stage 1: Tagraxofusp-erzs 9 µg/kg/da (N=3) | Stage 1: Tagraxofusp-erzs 12 µg/kg/Day (N=3) | Stage 2: Tagraxofusp-erzs 12 µg/kg/Day (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Irritable Bowel Syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Dysarthria (Psychiatric disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: Tagraxofusp-erzs 7 µg/kg/Day (N=3) | Stage 1: Tagraxofusp-erzs 9 µg/kg/da (N=3) | Stage 1: Tagraxofusp-erzs 12 µg/kg/Day (N=3) | Stage 2: Tagraxofusp-erzs 12 µg/kg/Day (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 3 | 3
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 2 | 3
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Retching (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Chest pain (General disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 3 | 2
Fatigue (General disorders) | 1 | 1 | 2 | 3
Oedema peripheral (General disorders) | 0 | 0 | 1 | 3
Pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 3 | 3
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 2 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 2 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0
Blood bilirubin (Investigations) | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 1
Blood urea increased (Investigations) | 0 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 1 | 0
Weight increased (Investigations) | 1 | 1 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 1
Headache (Nervous system disorders) | 1 | 1 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Dysarthria (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 1 | 1
Flushing (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The small number of patients treated at 12 µg/kg/day precluded definitive interpretation of the efficacy data from this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT02270463/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT02270463/SAP_001.pdf